CLINICAL TRIAL: NCT04718389
Title: A 52-week, Randomised, Double-blind, Double-dummy, Parallel Group, Multi-centre, Non-inferiority Study Assessing Exacerbation Rate, Additional Measures of Asthma Control and Safety in Adult and Adolescent Severe Asthmatic Participants With an Eosinophilic Phenotype Treated With GSK3511294 Compared With Mepolizumab or Benralizumab
Brief Title: A Study of GSK3511294 (Depemokimab) Compared With Mepolizumab or Benralizumab in Participants With Severe Asthma With an Eosinophilic Phenotype
Acronym: NIMBLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 206785
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Asthma
Keywords: Asthma; GSK3511294 (Depemokimab); Mepolizumab; Benralizumab; Interventional; Eosinophilic phenotype
MeSH Terms: conditions — Asthma | interventions — mepolizumab; benralizumab; Standard of Care

STUDY DESIGN:
Intervention Model Description: This is randomized, double-blind, parallel group, multi-center and non-inferiority study.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Participants receiving GSK3511294 (Depemokimab) plus placebo matching prior anti-IL-5/5R treatment (Experimental): Participants will receive GSK3511294 (Depemokimab) plus placebo treatment matching the active comparator (participant's anti-Interleukin-5/ 5 receptor [anti-IL-5/5R] treatment prior to randomization): either placebo matching mepolizumab or placebo matching benralizumab. All participants will continue their non-biologic Baseline SoC asthma treatment throughout the study.
  Interventions: Biological: GSK3511294 (Depemokimab); Biological: Placebo; Drug: Standard of care (SoC); Device: Pre-filled Syringes (PFS)
- Participants receiving prior anti-IL-5/5R treatment plus placebo matching GSK3511294 (Depemokimab) (Active Comparator): Participants will receive active comparator (participant's anti-IL-5/5R treatment prior to randomization): either mepolizumab or benralizumab, plus placebo matching GSK3511294 (Depemokimab). All participants will continue their non-biologic Baseline SoC asthma treatment throughout the study.
  Interventions: Biological: Mepolizumab; Biological: Benralizumab; Biological: Placebo; Drug: Standard of care (SoC); Device: Pre-filled Syringes (PFS)

INTERVENTIONS:
Biological: GSK3511294 (Depemokimab) — GSK3511294 (Depemokimab) will be provided in a single-use prefilled syringe (PFS).
  Arms: Participants receiving GSK3511294 (Depemokimab) plus placebo matching prior anti-IL-5/5R treatment
Biological: Mepolizumab — Mepolizumab will be provided in a single-use PFS.
  Arms: Participants receiving prior anti-IL-5/5R treatment plus placebo matching GSK3511294 (Depemokimab)
Biological: Benralizumab — Benralizumab will be provided in a single-use PFS.
  Arms: Participants receiving prior anti-IL-5/5R treatment plus placebo matching GSK3511294 (Depemokimab)
Biological: Placebo — Placebo will be a sterile liquid formulation.
Drug: Standard of care (SoC) — Non-biologic SoC will include inhaled corticosteroid (ICS) plus at least one other controller, long-acting beta-2-agonist (LABA), long-acting muscarinic antagonist (LAMA), with or without maintenance oral corticosteroids (OCS).
Device: Pre-filled Syringes (PFS) — PFS will include glass barrel with pre-staked needle and plunger.

SUMMARY:
This study will assess whether switching participants who have benefitted from mepolizumab or benralizumab to GSK3511294 (Depemokimab) is non-inferior to maintaining current treatment on the annualized rate of clinically significant exacerbations in participants with severe asthma with an eosinophilic phenotype. Throughout the study, all participants will continue their non-biologic Baseline standard of care (SoC) asthma treatment.

ELIGIBILITY:
Key inclusion criteria for study:

* Adult and adolescent participants more than or equal to (>=)12 years of age, at the time of signing the informed consent/assent.
* Participants who have a documented physician diagnosis of asthma for >=2 years that meets the National Heart, Lung, and Blood Institute guidelines (NHLBI) or Global Initiative for Asthma (GINA) guidelines.
* Participants receiving either mepolizumab 100 milligrams (mg) or benralizumab 30 mg for >=12 months prior to screening and have a documented benefit to therapy assessed by either:

  (i) >=50% reduction in exacerbation frequency since initiating treatment, or (ii) >=50% reduction in maintenance OCS use since initiating treatment, or (iii) No exacerbations in the past 6 months whilst receiving anti-IL-5/5R therapy and an Asthma Control Questionnaire (ACQ)-5 score of less than or equal to (<=)1.5 at screening.
* A well-documented requirement for regular treatment with medium to high dose ICS in the 12 months prior to Visit 1 with or without maintenance OCS. The maintenance ICS dose must be >=440 micrograms (mcg) fluticasone propionate (FP) hydrofluoroalkane (HFA) product daily, or clinically comparable. Participants who are treated with medium dose ICS will also need to be treated with a LABA to qualify for inclusion.
* Current treatment with at least one additional controller medication, besides ICS [for example (e.g.), LABA, LAMA, leukotriene receptor antagonist (LTRA), or theophylline].

Key exclusion criteria for study:

* Participants with presence of a known pre-existing, clinically important lung condition other than asthma. This includes (but is not limited to) current infection, bronchiectasis, pulmonary fibrosis, bronchopulmonary aspergillosis, or diagnoses of emphysema or chronic bronchitis (chronic obstructive pulmonary disease other than asthma) or a history of lung cancer.
* Participants with other conditions that could lead to elevated eosinophils such as hyper-eosinophilic syndromes including (but not limited to) Eosinophilic Granulomatosis with Polyangiitis (EGPA, formerly known as Churg-Strauss Syndrome) or Eosinophilic Esophagitis.
* A current malignancy or previous history of cancer in remission for less than 12 months prior to screening (Participants that had localized carcinoma of the skin which was resected for cure will not be excluded).
* Cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice.
* Participants with current diagnosis of vasculitis. Participants with high clinical suspicion of vasculitis at screening will be evaluated and current vasculitis excluded prior to enrolment.
* Participants who have received Omalizumab (Xolair), dupilumab (Dupixent) or reslizumab (Cinqair/Cinqaero) within 130 days prior to Visit 1.
* Participants who have received any Monoclonal antibody (mAb) within 5 half-lives of Visit 1.
* Corrected QT interval using Fridericia's formula (QTcF) >=450 milliseconds (msec) or QTcF >=480 msec for participants with Bundle Branch Block at screening Visit 1.
* Current smokers or former smokers with a smoking history of >=10 pack years (number of pack years equal to [number of cigarettes per day/20] times number of years smoked). A former smoker is defined as a participant who quit smoking at least 6 months prior to Visit 1.
* Participants with allergy/intolerance to a mAb or biologic.

Key exclusion criteria for randomization:

* Evidence of a clinically significant abnormality in the 12-lead electrocardiogram (ECG) over-read conducted at Screening Visit 1, based on the evaluation of the investigator, or QTcF >=450 msec or QTcF >=480 msec for participants with Bundle Branch Block, at randomization Visit 2.
* Participants with a clinically significant asthma exacerbation in the 7 days prior to randomization should have their randomization visit delayed until the investigator considers the participant's asthma to be stable. If the 8-week screening period has elapsed, then the participant should be considered a run-in failure.
* Any changes in the dose or regimen of Baseline ICS and/or additional controller medication (except for treatment of an exacerbation) during the run-in period.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1719 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2025-09-14 (Actual); Study Completion 2025-09-14 (Actual)

PRIMARY OUTCOMES:
Annualized rate of clinically significant exacerbations over 52 weeks | Up to Week 52
  Clinically significant exacerbations of asthma are defined by worsening of asthma which requires use of systemic corticosteroids and/or hospitalization and/or Emergency Department (ED) visit. Annualized rate of exacerbations will be calculated as number of exacerbations experienced by the participant divided by the length of time the participant is measured on.

SECONDARY OUTCOMES:
Weighted mean change from Baseline in St. George's Respiratory Questionnaire (SGRQ) total score | Baseline (Day 1) and up to Week 52
  The SGRQ is a well-established instrument, comprising 51 questions designed to measure Quality of Life in participants with diseases of airway obstruction. Higher score indicates worse quality of life.
Weighted mean change from Baseline in Asthma Control Questionnaire-5 (ACQ-5) score | Baseline (Day 1) and up to Week 52
  The ACQ-5 is a five-item questionnaire, which has been developed as a measure of participants' asthma control that can be quickly and easily completed. The five questions enquire about the frequency and/or severity of symptoms (nocturnal awakening on waking in the morning, activity limitation, and shortness of breath, wheeze) over the previous week. The response options for all these questions consist of a zero (no impairment/limitation) to six (total impairment/ limitation) scale. Higher score indicates more limitations.
Weighted mean change from Baseline in pre-bronchodilator forced expiratory volume in one second (FEV1) | Baseline (Day 1) and up to Week 52
  FEV1 is a measure of pulmonary function and is the maximum amount of air that can be forced out in one second after taking a deep breath. FEV1 will be measured using spirometry.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (307):
- United States (97):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Scottsboro, Alabama
  - GSK Investigational Site, Litchfield Park, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Encinitas, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Oxnard, California
  - GSK Investigational Site, Rancho Cucamonga, California
  - GSK Investigational Site, Redondo Beach, California
  - GSK Investigational Site, Redwood City, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Valencia, California
  - GSK Investigational Site, Woodland, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Kissimmee, Florida
  - GSK Investigational Site, Loxahatchee Groves, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Lakes, Florida
  - GSK Investigational Site, North Palm Beach, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Sebring, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Calhoun, Georgia
  - GSK Investigational Site, Glenview, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Bangor, Maine
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Chevy Chase, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Burlington, Massachusetts
  - GSK Investigational Site, New Bedford, Massachusetts
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Flint, Michigan
  - GSK Investigational Site, Warren, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Gulfport, Mississippi
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Brick, New Jersey
  - GSK Investigational Site, Northfield, New Jersey
  - GSK Investigational Site, Riverdale, New Jersey
  - GSK Investigational Site, Toms River, New Jersey
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Corning, New York
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Huntersville, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Corvallis, Oregon
  - GSK Investigational Site, Altoona, Pennsylvania
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Wyomissing, Pennsylvania
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Hendersonville, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Amarillo, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Kerrville, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Williamsburg, Virginia
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Greenfield, Wisconsin
- Australia (16):
  - GSK Investigational Site, Macquarie Park, New South Wales
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Cairns, Queensland
  - GSK Investigational Site, South Brisbane, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Bedford Park, South Australia
  - GSK Investigational Site, North Adelaide, South Australia
  - GSK Investigational Site, Toorak Gardens, South Australia
  - GSK Investigational Site, Woodville, South Australia
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Fitzroy, Victoria
  - GSK Investigational Site, Frankston, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Austria (2):
  - GSK Investigational Site, Feldbach
  - GSK Investigational Site, Vienna
- Canada (10):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Moncton, New Brunswick
  - GSK Investigational Site, Ajax, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- Finland (2):
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- France (26):
  - GSK Investigational Site, Amiens
  - GSK Investigational Site, Annecy
  - GSK Investigational Site, Antony
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Cannes
  - GSK Investigational Site, Cholet
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, La Tronche
  - GSK Investigational Site, Le Mans
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montfermeil
  - GSK Investigational Site, Montivilliers
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pontoise
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Saint-Herblain
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Suresnes
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Tours
- Germany (20):
  - GSK Investigational Site, Aschaffenburg
  - GSK Investigational Site, Bendorf
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Bonn
  - GSK Investigational Site, Darmstadt
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Fürstenwalde
  - GSK Investigational Site, Geesthacht
  - GSK Investigational Site, Halle
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Hanover
  - GSK Investigational Site, Landsberg
  - GSK Investigational Site, Leipzig
  - GSK Investigational Site, Lübeck
  - GSK Investigational Site, Magdeburg
  - GSK Investigational Site, Mainz
  - GSK Investigational Site, München
  - GSK Investigational Site, Neu-Isenburg
  - GSK Investigational Site, Rheine
  - GSK Investigational Site, Schleswig
- Ireland (2):
  - GSK Investigational Site, Cork
  - GSK Investigational Site, Dublin
- Israel (8):
  - GSK Investigational Site, Beersheba
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Tel Aviv
  - GSK Investigational Site, Zrifin
- Italy (28):
  - GSK Investigational Site, Bari
  - GSK Investigational Site, Bergamo
  - GSK Investigational Site, Bologna
  - GSK Investigational Site, Brescia
  - GSK Investigational Site, Catania
  - GSK Investigational Site, Ferrara
  - GSK Investigational Site, Florence
  - GSK Investigational Site, Genova
  - GSK Investigational Site, Mantova
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Modena
  - GSK Investigational Site, Monserrato CA
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Padua
  - GSK Investigational Site, Palermo
  - GSK Investigational Site, Pavia
  - GSK Investigational Site, Perugia
  - GSK Investigational Site, Pisa
  - GSK Investigational Site, Reggio Emilia
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Salerno
  - GSK Investigational Site, Sassari
  - GSK Investigational Site, Siena
  - GSK Investigational Site, Torino
  - GSK Investigational Site, Torrette AN
  - GSK Investigational Site, Treviso
  - GSK Investigational Site, Trieste
  - GSK Investigational Site, Verona
- Japan (27):
  - GSK Investigational Site, Shibuya-Ku, Tokyo
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Akita
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Fukushima
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Numakunai
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shimane
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Toyama
  - GSK Investigational Site, Wakayama
- Netherlands (10):
  - GSK Investigational Site, Arnhem
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Deventer
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Harderwijk
  - GSK Investigational Site, Leeuwarden
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Zwolle
- Norway (2):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Lrenskog
- Portugal (4):
  - GSK Investigational Site, Coimbra
  - GSK Investigational Site, Guarda
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Matosinhos Municipality
- GSK Investigational Site, Guaynabo, Puerto Rico
- GSK Investigational Site, Golnik, Slovenia
- Spain (21):
  - GSK Investigational Site, Alcorcón
  - GSK Investigational Site, Almería
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Benalmádena
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Jerez de la Frontera
  - GSK Investigational Site, La Laguna Santa Cruz
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, MErida Badajoz
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Pozuelo de AlarcOn Madr
  - GSK Investigational Site, Salamanca
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Via-Real CastellOn
  - GSK Investigational Site, Vitoria-Gasteiz
  - GSK Investigational Site, Zaragoza
- Sweden (5):
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Östersund
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
- Switzerland (4):
  - GSK Investigational Site, Aarau
  - GSK Investigational Site, Basel
  - GSK Investigational Site, Liestal
  - GSK Investigational Site, Sankt Gallen
- Taiwan (5):
  - GSK Investigational Site, Banchiau Taipei
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Linkou - Taoyuan Hsien
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
- United Kingdom (16):
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Bristol Avon
  - GSK Investigational Site, Cottingham
  - GSK Investigational Site, Exeter
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Portsmouth
  - GSK Investigational Site, Preston
  - GSK Investigational Site, Wakefield
  - GSK Investigational Site, Wishaw

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com